CLINICAL TRIAL: NCT06004947
Title: An Open-Label, Phase 1 Study in Healthy Volunteers to Evaluate the Drug-Drug Interaction Potential of CCX168 With Concomitant Medications
Brief Title: A Study in Healthy Volunteers to Evaluate the Drug-Drug Interaction Potential of CCX168 With Concomitant Medications
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: CL008_168
Record Dates: First submitted 2023-08-15; First posted 2023-08-22 (Actual); Last update posted 2023-08-22 (Actual); Status verified 2023-08

CONDITIONS: Anti-neutrophil Cytoplasmic Antibody-associated Vasculitis
Keywords: Renal diseases; Atypical hemolytic uremic syndrome; Immunoglobulin A nephropathy; Complement 5a receptor (C5aR); Complement
MeSH Terms: conditions — Anti-Neutrophil Cytoplasmic Antibody-Associated Vasculitis; Kidney Diseases; Atypical Hemolytic Uremic Syndrome; Glomerulonephritis, IGA | interventions — avacopan; Midazolam; Celecoxib; Itraconazole; Rifampin

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cohort A (Experimental): A single dose of 2 mg midazolam (a Cytochrome P450 [CYP]3A4 probe drug) and a single dose of 200 mg celecoxib (a CYP2C9 probe drug) will be given orally concurrently on Day 1 and Day 13. On Day 3 through Day 18, CCX168 will be given orally at 30 mg twice daily (b.i.d.), and a single dose of 30 mg CCX168 will be given in the morning on Day 19. On Day 16 through Day 19, a once daily (q.d.) dose of 200 mg itraconazole (a CYP3A4 inhibitor) will be given orally.
  Interventions: Drug: CCX168; Drug: Midazolam; Drug: Celecoxib; Drug: Itraconazole
- Cohort B (Experimental): A single dose of 30 mg CCX168 will be given on Day 1 and Day 14, while rifampicin (a CYP3A4 inducer) will be given at 600 mg once daily from Day 4 through Day 17.
  Interventions: Drug: CCX168; Drug: Rifampicin

INTERVENTIONS:
Drug: CCX168 — Administered orally.
Drug: Midazolam — Administered orally.
  Arms: Cohort A
Drug: Celecoxib — Administered orally.
  Arms: Cohort A
Drug: Itraconazole — Administered orally.
  Arms: Cohort A
Drug: Rifampicin — Administered orally.
  Arms: Cohort B

SUMMARY:
The primary objective of this study will be to evaluate the drug-drug interaction potential of CCX168 with concomitant medications, as either a perpetrator or a victim, following oral administration of CCX168 to healthy participants.

ELIGIBILITY:
Inclusion Criteria:

* Male or female participants, aged 18-55 years inclusive, who are in generally good health as judged by the Investigator, whose body mass index is 19.0 to 32.0 kg/m^2 inclusive;
* Willing and able to give written Informed Consent and to comply with the requirements of the study protocol;
* Negative result of the human immunodeficiency virus screen, the hepatitis B screen, and the hepatitis C screen;
* Judged to be healthy by the Investigator, based on medical history, physical examination (including electrocardiogram, and clinical laboratory assessments. Participants with clinical laboratory values that are outside of normal limits and/or with other abnormal clinical findings that are judged by the Investigator not to be of clinical significance may be entered into the study;
* Female participants of childbearing potential, or male participants with partners of childbearing potential may participate if adequate contraception is used during, and for at least 90 days after, any administration of study medication.

Exclusion Criteria:

* Pregnant or breastfeeding;
* Used a prescription and/or over-the-counter medication, with the exception of ibuprofen, hormonal contraceptives, and multi-vitamins, within 14 days prior to check-in; herbal supplements must be stopped 7 days prior to check-in;
* For at least 14 days prior to check-in and throughout the blood sample collection period, participants will not be allowed to eat any food or drink any beverage containing alcohol, grapefruit or grapefruit juice, apple or orange juice, vegetables from the mustard green family (e.g., kale, broccoli, watercress, collard greens, kohlrabi, Brussels sprouts, mustard greens) and charbroiled meats; strenuous exercise must be stopped 4 days prior to check-in;
* History within the three months prior to check-in of use of tobacco and/or nicotine containing products;
* History within one year prior to check-in of illicit drug use;
* History of alcohol abuse at any time in the past;
* Has a history or presence of any form of cancer within the 5 years prior to check-in, with the exception of excised basal cell or squamous cell carcinoma of the skin, or cervical carcinoma in situ or breast carcinoma in situ that has been excised or resected completely and is without evidence of local recurrence or metastasis;
* History or presence of unexplained syncope or family history of sudden death, or any medical condition or disease which, in the opinion of the Investigator, may place the participant at unacceptable risk for study participation;
* Donated or lost more than 350 mL of blood or blood products within 56 days prior to screening, or donated plasma within 7 days of dosing;
* Participant's hemoglobin less than 11.5 g/dL for women or less than 13.0 g/dL for men, at screening or check-in, confirmed by a repeat measurement;
* Participated in any clinical study of an investigational product within 30 days prior to dosing or within 5 half-lives after dosing;
* Participant has any evidence of hepatic disease; aspartate aminotransferase, alanine aminotransferase, alkaline phosphatase, or bilirubin greater than 1.5 times the upper limit of normal at screening or check-in;
* Participant's white blood cell count is below the lower limit of normal at screening or check-in, confirmed by a repeat measurement;
* Participant has any evidence of renal impairment; serum creatinine greater than 1.5 times the upper limit of normal at screening or check-in;
* Participant's urine tested positive at screening and/or check-in for any of the following: opioids, amphetamines and methamphetamines, cannabinoids, benzodiazepines, barbiturates, cocaine, cotinine, methylenedioxymethamphetamine (MDMA or "ecstasy"), methadone, phencyclidine, tri-cyclic antidepressants, or alcohol (Breathalyzer test allowed for alcohol).
* Participant is known as a CYP2C9 poor metabolizer.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2016-01-14 (Actual); Primary Completion 2016-03-15 (Actual); Study Completion 2016-06-10 (Actual)

PRIMARY OUTCOMES:
Cohort A: Maximum Plasma Concentration (Cmax) of Midazolam | Up to Day 13
Cohort A: Cmax of Celecoxib | Up to Day 13
Cohort A: Time of Cmax (Tmax) of Midazolam | Up to Day 13
Cohort A: Tmax of Celecoxib | Up to Day 13
Cohort A: Area under the plasma concentration-time curve (AUC) from Time 0 to infinity of Midazolam | Up to Day 13
Cohort A: AUC from Time 0 to infinity of Celecoxib | Up to Day 13
Cohort A: Apparent Terminal Half Life of Midazolam | Up to Day 13
Cohort A: Apparent Terminal Half Life of Celecoxib | Up to Day 13
Cohort A: Cmax of CCX168 | Day 15 up to Day 19
Cohort A: Tmax of CCX168 | Day 15 up to Day 19
Cohort A: AUC Over the Dosing Interval of CCX168 | Day 15 up to Day 19
Cohort B: Cmax of CCX168 | Up to Day 14
Cohort B: Tmax of CCX168 | Up to Day 14
Cohort B: AUC from Time 0 to infinity of CCX168 | Up to Day 14
Cohort B: Apparent Terminal Half Life of CCX168 | Up to Day 14

SECONDARY OUTCOMES:
Number of Participants Experiencing Adverse Events (AEs) | Up to Day 29
Number of Participants Experiencing Clinically Significant Changes in Laboratory Parameters | Up to Day 19
Number of Participants Experiencing Clinically Significant Changes in Vital Sign Parameters | Up to Day 19

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (1):
- Celerion, Tempe, Arizona, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data sharing requests relating to this study will be considered beginning 18 months after the study has ended and either 1) the product and indication have been granted marketing authorization in both the US and Europe or 2) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this study.
Access Criteria: Qualified researchers may submit a request containing the research objectives, the Amgen product(s) and Amgen study/studies in scope, endpoints/outcomes of interest, statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). In general, Amgen does not grant external requests for individual patient data for the purpose of re-evaluating safety and efficacy issues already addressed in the product labelling. Requests are reviewed by a committee of internal advisors. If not approved, a Data Sharing Independent Review Panel will arbitrate and make the final decision. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement. This may include anonymized individual patient data and/or available supporting documents, containing fragments of analysis code where provided in analysis specifications. Further details are available at the URL below.
URL: http://www.amgen.com/datasharing

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com